CLINICAL TRIAL: NCT02698930
Title: Effect of Dexmedetomidine on Postoperative Renal Function in Infective Endocarditis Patients Undergoing Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2015-0839
Record Dates: First submitted 2016-02-15; First posted 2016-03-04 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; acute kidney injury; dexmedetomidine
MeSH Terms: conditions — Endocarditis; Acute Kidney Injury | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine group (Experimental)
  Interventions: Drug: dexmedetomidine
- Control group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: dexmedetomidine — Randomly selected patients of the dexmedetomidine group are given intravenous 0.4mcg/kg/h of dexmedetomidine from the beginning of the anesthesia to postoperative 1 day.
  Arms: dexmedetomidine group
Drug: Normal saline — Group given intravenous 0.4mcg/kg/h of normal saline from the beginning of the anesthesia to postoperative 1 day.
  Arms: Control group

SUMMARY:
Acute kidney injury is major complication after open heart surgery. The cause of acute kidney injury following open heart surgery is related to activation of sympathetic nervous system, decrease of renal blood flow, ischemia-reperfusion injury and systemic inflammatory response.

Infective endocarditis patients undergoing open heart surgery have systemic inflammatory response associated with infective endocarditis. And the inflammatory response can be aggravated by cardiopulmonary bypass. The incidence of acute kidney injury following open heart surgery due to infective endocarditis was 50% in a previous report. And this acute kidney injury was related to the poor outcome and high mortality. Thus, the preventive method to protect kidney function will be needed in the patients with infective endocarditis undergoing open heart surgery.

Dexmedetomidine is a selective α2-agonist and has sedative, analgesic, and CNS depressive effect. And several experimental study demonstrated the renal protective effect. Intraoperative dexmedetomidine administration can reduce the amount of anesthetics needed and suppress the sympathetic response resulted by surgical stimulation. And dexmedetomidine was reported to reduce the level of serum cortisol, epinephrine and norepinephrine during the operation. Thus, these effects of dexmedetomidine can be expected to reduce the incidence of acute kidney injury.

Therefore, the investigators hypothesized that dexmedetomidine has renal protective effect and this effect might be related to the suppression of inflammatory response. Thus, the investigators will evaluate the incidence of acute kidney injury and the incidence of major adverse kidney events (MAKE) after open heart surgery due to infective endocarditis and the level of inflammatory mediators.

The primary end point of this study is the incidence of acute kidney injury after open heart surgery due to infective endocarditis. And secondary end point is the incidence of MAKE, the level of cystatin C which is related to the renal function, the level of inflammatory mediator and the postoperative morbidities.

ELIGIBILITY:
Inclusion Criteria:

* patients with infective endocarditis
* patients who are scheduled to undergo open heart surgery

Exclusion Criteria:

* chronic kidney disease
* taking high dose steroid (>10mg/day prednisolone or equivalent)
* age under 20 years
* cognitive dysfunction
* disabling mental change disorder
* unable to communicate or speak Korean

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of acute kidney injury | 1 week

SECONDARY OUTCOMES:
Cystatin C level | postoperative day 1,2,3 and 5
  serum cystatin C level (mg/L)
inflammatory mediator(IL-6) level | postoperative day 1,2,3 and 5
  serum inflammatory mediator (IL-6(pg/mL)
inflammatory mediator(CRP) level | postoperative day 1,2,3 and 5
  serum inflammatory mediator (CRP(mg/L))
inflammatory mediator(WBC) level | postoperative day 1,2,3 and 5
  Serum WBC(/microL) level
inflammatory mediator(neutrophil count) level | postoperative day 1,2,3 and 5
  serum inflammatory mediator (neutrophil count(/microL)) level
serum norepinephrine/epinephrine level(ng/mL) | postoperative day 1,2,3 and 5
intraoperative hemodynamics measured by amount of used vasopressors(mL) | postoperative day 1,2,3 and 5
intraoperative fluid intake and output | postoperative day 1,2,3 and 5
  intraoperative intake and output measured by the amount of fluid(crystalloid/colloid)(mL) and blood administered(mL)
postoperative complications | postoperative day 1,2,3 and 5
  postoperative complications such as development of myocardial infarction, arrhythmia, cerebrovascular accident, wound infection, and mortality.
Major adverse kidney events (MAKE) | 3month, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosner MH, Portilla D, Okusa MD. Cardiac surgery as a cause of acute kidney injury: pathogenesis and potential therapies. J Intensive Care Med. 2008 Jan-Feb;23(1):3-18. doi: 10.1177/0885066607309998. PMID 18230632
- [Background] Conlon PJ, Jefferies F, Krigman HR, Corey GR, Sexton DJ, Abramson MA. Predictors of prognosis and risk of acute renal failure in bacterial endocarditis. Clin Nephrol. 1998 Feb;49(2):96-101. PMID 9524779
- [Background] Ren J, Zhang H, Huang L, Liu Y, Liu F, Dong Z. Protective effect of dexmedetomidine in coronary artery bypass grafting surgery. Exp Ther Med. 2013 Aug;6(2):497-502. doi: 10.3892/etm.2013.1183. Epub 2013 Jun 25. PMID 24137215